CLINICAL TRIAL: NCT06157918
Title: A Single-Center, Randomized, Open-label, Single-dose, 3-Sequence, 3-Period Rossover Design to Evaluate the Relative Bioavailability and Food Effect of SYHA1813 Oral Solution in Healthy Participants
Brief Title: Relative Bioavailability and Food Effect of SYHA1813 Oral Solution in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Runshi Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SYHA1814-003
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Intervention Model Description: 3-period Crossover Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1-sequence ABC (Experimental): Participants will sequentially receive SYHA1813 oral solution (2.0g:25mg) fasted (Treatment A), followed by SYHA1813 oral solution (20ml:200mg) fasted (Treatment B), and SYHA1813 oral solution (2.0g:25mg) fed (Treatment C).
  Interventions: Drug: SYHA1813 oral solution (2.0g:25mg); Drug: SYHA1813 oral solution (20ml:200mg)
- Group 2-sequence BCA (Experimental): Participants will sequentially receive SYHA1813 oral solution (20ml:200mg) fasted (Treatment B), followed by SYHA1813 oral solution (2.0g:25mg) fed(Treatment C), and SYHA1813 oral solution (2.0g:25mg) fasted (Treatment A).
  Interventions: Drug: SYHA1813 oral solution (2.0g:25mg); Drug: SYHA1813 oral solution (20ml:200mg)
- Group 3-sequence CAB (Experimental): Participants will sequentially receive SYHA1813 oral solution (2.0g:25mg) fed (Treatment C), followed by SYHA1813 oral solution (2.0g:25mg) fasted (Treatment A), and SYHA1813 oral solution (20ml:200mg) fasted (Treatment B).
  Interventions: Drug: SYHA1813 oral solution (2.0g:25mg); Drug: SYHA1813 oral solution (20ml:200mg)

INTERVENTIONS:
Drug: SYHA1813 oral solution (2.0g:25mg) — SYHA1813 oral solution, 25mg, oral
Drug: SYHA1813 oral solution (20ml:200mg) — SYHA1813 oral solution, 25mg, oral

SUMMARY:
This is a three-period crossover phase I study designed to evaluate the relative bioavailability, food effect, safety and tolerability of SYHA1813 oral solution in healthy participants.

DETAILED DESCRIPTION:
Avoid duplicating information that will be entered elsewhere, such as Eligibility Criteria or Outcome Measures.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male aged 18 to 60 years old;
2. Weight more than 50.0 kg and body mass index between 19 to 26.0 kg/m^2;
3. Normal or abnormal results without clinical significance on all tests including medical history, vital signs, physical examination, laboratory evaluation (routine blood, blood biochemistry, urine routine, coagulation function, serum virology, and other related tests), 12-lead electrocardiogram, chest X-ray and other tests;
4. Male participants and their partners must agree to use effective non-hormonal contraception from the first administration of the test drug to 6 months after the last administration of the test drug, even if permanent contraception has already been used, and the male participant does not plan to donate sperm;
5. Voluntarily sign the informed consent form, and cooperate in completing the trial according to the protocol.

Exclusion Criteria:

1. Allergic constitution (allergic to 2 or more kinds of drugs, food, or pollen);
2. Participants with a clear history of neurological disease or psychiatric disease, a history of severe cardiovascular, hepatic, renal, endocrine, respiratory, hematologic, digestive, immune, and other various systemic diseases, or a history of malignant neoplastic disease;
3. Participants who are unable to swallow orally administered drugs, or clinically significant abnormalities in gastrointestinal function that could affect drug absorption, distribution, metabolism, and excretion;
4. Participants who have undergone major surgery within 6 months prior to screening or who are scheduled to undergo surgery during the trial;
5. Participants with 1 or more abnormal vital signs at screening;
6. Abnormal and clinically significant electrocardiograms: QTc interval >450ms;
7. Participants who consumed more than 14 units of alcohol per week in the 4 weeks prior to screening or who had a positive breath test for alcohol at screening;
8. Smoking ≥ 5 cigarettes per day on average within 6 months prior to screening;
9. Participants with a history of drug or substance abuse, or a positive urine drug screen;
10. Participants who have lost blood or donated more than 400 ml of blood within 4 weeks prior to screening or plan to donate blood during the study or within 1 month of the end of the study;
11. Participants who have participated in other clinical trials within 3 months prior to screening;
12. Habitual intake of excessive xanthine or caffeine-containing foods, beverages, or other foods that interfere with drug absorption, distribution, metabolism, excretion within 4 weeks prior to screening;
13. Participants who have taken a special diet (dragon fruit, mango, grapefruit, lime, poppy seed, or food or drink prepared from them) within 7 days prior to screening, or participants who are unable to stop taking the above special diets during the trial;
14. Participants who have used potent inhibitors or inducers of CYP enzymes (e.g., CYP2C9, 2C19, and 3A4) within 4 weeks prior to screening;
15. Participants who have used prescription, over-the-counter, herbal, vitamin, or mineral medications within 2 weeks prior to screening, and participants who have taken medications prior to screening that have not completed 5 half-lives, whichever is longer among the various medications;
16. Participants who cannot tolerate venipuncture or with a history of fainting needle or blood;
17. Participants who are lactose intolerant;
18. Any condition that the investigator considers inappropriate for participation in the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 19 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Cmax | Up to 120 hours post-dose for eachperiod
  Maximum observed plasma concentration
AUC0-∞ | Up to 120 hours post-dose for eachperiod
  Area under the plasma concentration time curve from time zero extrapolated to infinite time
AUC0-t | Up to 120 hours post-dose for eachperiod
  Area under the plasma concentration time curve from time zero to the time of the last quantifiable concentration

SECONDARY OUTCOMES:
Tmax | Up to 120 hours post-dose for eachperiod
  Time of maximum observed plasma concentration
T1/2 | Up to 120 hours post-dose for eachperiod
  Terminal elimination half-life
Title:Cl/F | Up to 120 hours post-dose for eachperiod
  Apparent total body clearance
V/F | Up to 120 hours post-dose for eachperiod
  Apparent volume of distribution
Number of participants with Adverse Events | Up to 34 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Shanghai, China

IPD SHARING:
Plan to Share IPD: No